CLINICAL TRIAL: NCT06728189
Title: A Clinical Research Evaluating the Safety and Efficacy of CD70-targeted CAR-NKT Cells (CGC738) Therapy in Subjects with Advanced Malignant Solid Tumors
Brief Title: A Clinical Research About CD70-targeted CAR-NKT Cells Therapy in Subjects with Advanced Malignant Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Collaborators: Suzhou Cure Genetics Biosciences Co., Limited. (Unknown)
Responsible Party: Principal Investigator, Jun Guo, Deputy Director of Peking University Cancer Hospital & Institute；Director of Renal Cancer and Melanoma Department., Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CGC738-IIT-01
Record Dates: First submitted 2024-11-22; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Advanced Malignant Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CAR-NKT Cells Lymphodepleting regimen (Experimental): Cyclophosphamide + Fludarabine + Infusion of CAR-NKT Cells Lymphodepleting regimen, Cyclophosphamide 250mg/m2 IV on day -5 to -3 and Fludarabine 25mg/m2 IV on days -5 to -3. Followed by infusion of CAR-NKT on day 0.
  Interventions: Biological: CAR-NKT Cells treatment

INTERVENTIONS:
Biological: CAR-NKT Cells treatment — Cyclophosphamide + Fludarabine + Infusion of CAR-NKT Cells Lymphodepleting regimen, Cyclophosphamide 250mg/m2 IV on day -5 to -3 and Fludarabine 25mg/m2 IV on days -5 to -3. Followed by infusion of CAR-NKT on day 0.
  Potential CGC738 doses:
  Dose level 1: 5.0×106 CAR- NKT cells/m2; Dose level 2: 1.5×107 CAR- NKT cells/m2; Dose level 3: 4.5×107 CAR- NKT cells/m2;

SUMMARY:
This is a phase I, open-label, single-arm study conducted to evaluate the efficacy, safety and PK of CGC738 in the treatment of advanced malignant solid tumors.

Condition or disease：advanced malignant solid tumors Intervention/treatment：Biological: CD70 CAR-NKT cells Phase：Phase 1

DETAILED DESCRIPTION:
This was a dose-expansion study, we plan to enroll 13 to 23 patients with CD70-positive advanced malignant solid tumors to CGC738 treatment. The study was conducted in two stages: dose escalation and dose expansion. Dose escalation involved three dose groups, which were administered using a rapid titration approach combined with the "3+3" design. Revised sentence: "One subject will be enrolled in the initial dose group, and if no dose-limiting toxicity (DLT) occurs within 28 days of the first administration, three additional subjects will be recruited into the subsequent predetermined escalating dose group. A particular dose level will be expanded to 6 patients if one patient out of 3 patients treated at that particular dose level develops DLT. Once this occurs, further dose-escalations are halted until the dose has proven to be safe in the expanded cohort. If 2 or more in a cohort of 6 patients develop DLT no further dose escalation is allowed, and the next lower dose level will be expanded to 6 patients in total. The highest dose among the dose levels tested at which no more than one out of six patients experiences DLT will be considered the MTD. Dose exploration can be discontinued once one or more dose levels with an acceptable safety profile and satisfactory antitumor activity have been selected for subsequent evaluation. During the treatment period of the study, three dose levels of CGC738 will be evaluated. Each of the dose levels will evaluate the safety of the CAR-NKT cells.

The extended study is anticipated to enroll a cohort of 6 to 10 participants. We used leukapheresis for cell collection. The lymphodepletion procedure was conducted using a combination of fludarabine and cyclophosphamide.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years.
2. ECOG 0-1 points.
3. The expected survival time is more than 3 months.
4. Patients with advanced advanced malignant solid tumor confirmed by histology or cytology to be recurrent or metastatic after at least second-line treatment.
5. IHC: CD70 positive.
6. At least one measurable lesion at baseline per RECIST version 1.1.
7. The functions of important organs are basically normal:
8. Pregnancy tests for women of childbearing age shall be negative, Both men and women agreed to use effective contraception.
9. Subjects or their guardians agree to participate in this clinical trial and sign the ICF, indicating that they understand the purpose and procedures of this clinical trial and are willing to participate in the research.

Exclusion Criteria:

1. Use of cell therapy within the previous one month.
2. Subjects with other malignant tumors within the past 2 years, except basal or squamous skin cancer, superficial bladder cancer, and breast cancer in situ, have been completely cured and do not need follow-up treatment.
3. Patients with leptomeningeal metastasis or central nervous system metastasis, and definite central nervous system underlying diseases with significant symptoms.
4. Immunotherapy, targeted drug therapy or chemotherapy within 5 drug half-lives within 2 weeks before cell infusion.
5. Active hepatitis B, HIV positive and HCV positive.
6. Active infection or uncontrollable infection.
7. Subjects with NYHA heart failure class ≥2 or hypertension uncontrolled by standard therapy requiring special treatment, previous history of myocarditis, or myocardial infarction within 6 months.
8. Unstable respiratory diseases, including interstitial pneumonia.
9. Uncontrolled ascites and pleural effusion
10. Known to have active or uncontrolled autoimmune diseases, such as Crohns disease, rheumatoid arthritis, systemic lupus erythematosus, etc. .
11. Subjects who are using systemic steroids or steroid inhalers for treatment.
12. Pregnant or lactating female subjects.
13. Other investigators deem it unsuitable to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2026-10-17 (Estimated); Study Completion 2026-10-17 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Experiencing Dose Limiting Toxicities (DLTs) | Day 28 after CGC738 infusion
  Dose limiting toxicity (DLT) is an AE that meets the following criteria and occurs within 28 days of CGC729 infusion.AE is graded according to CTCAE version 5.0.

SECONDARY OUTCOMES:
Assess Objective response rate (ORR) | Day 1 through week 56
Assess Disease control rate (DCR) | Day 1 through week 56
Incidence of adverse events (AEs) | Day 1 through week 56
Cmax, Tmax, AUCS of CD70 CAR-NKT cell dynamics | Day 1 through week 56

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No